CLINICAL TRIAL: NCT06310785
Title: Opioid-Free Anesthesia Utilizing Esketamine for Thoracoscopic Pulmonary Nodule Surgery: A Randomized Controlled Clinical Trial
Brief Title: Esketamine Anesthesia in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui Xu (Other)
Responsible Party: Sponsor-Investigator, Hui Xu, professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJ-IRB20231191
Record Dates: First submitted 2024-01-31; First posted 2024-03-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: General Anesthesia; Thoracic Surgery
MeSH Terms: interventions — Esketamine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Neither the patients who participated in the trial nor the analysis of the results of the study were aware of the experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): Patients in the esketamine group was induced with esketamine 0.5 mg/kg, propofol 2 mg/kg, and rocuronium 0.9 mg/kg. Anesthesia is maintained with propofol 5 mg/kg/h and esketamine 0.5 mg/kg/h
  Interventions: Drug: Esketamine
- opioid group (Active Comparator): Patients in the opioid group was induced with sufentanil 0.5 ug/kg, propofol 2 mg/kg, rocuronium 0.9 mg/kg. Anesthesia is maintained with propofol 5 mg/kg/h and remifentanil 0.1 ug/kg/min
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Esketamine — The esketamine group used esketamine as an analgesic during induction and maintenance of anesthesia.
  Arms: Esketamine group
Drug: Sufentanil — In the opioid group, sufentanil was used as an analgesic during anesthesia induction and remifentanil was used as an analgesic during anesthesia maintenance.
  Arms: opioid group

SUMMARY:
Patients in the esketamine group was induced with esketamine 0.5 mg/kg, propofol 2 mg/kg, and rocuronium 0.9 mg/kg. Anesthesia is maintained with propofol 5 mg/kg/h and esketamine 0.5 mg/kg/h. Patients in the opioid group was induced with sufentanil 0.5 ug/kg, propofol 2 mg/kg, rocuronium 0.9 mg/kg. Anesthesia is maintained with propofol 5 mg/ kg/h and remifentanil 0.1 ug/kg/min.

DETAILED DESCRIPTION:
Before anesthesia induction, radial artery puncture and catheterization under local anesthesia for manometry, and intravenous dexmedetomidine (1 µg/kg) infused over 15 minutes, followed by penehyclidine hydrochloride (0.01mg/kg), palonosetron (0.075 mg), dexamethasone (5 mg). Anesthesia-induced in the opioid group (group A) was intravenous sufentanil 0.5 ug/kg, and esketamine group (group E) received intravenous esketamine 0.5 mg/kg. Subsequently, both groups were sequentially injected with propofol 2 mg/kg and rocuronium 0.9 mg/kg. After the onset of rocuronium, the left-sided double-lumen endotracheal tube was guided by a video laryngoscope, the correct position of the tube was confirmed by bronchoscope, and the anesthesia machine was connected to the tube for mechanical ventilation after fixation, with a tidal volume of 6-8 mL/kg (ideal body weight), a respiratory rate of 10~18 breaths/min, and end-expiratory carbon dioxide partial pressure at 35~45 mmHg (4.7-6.0 kPa).

Intraoperative anesthesia maintenance in the opioid group was pumped with propofol (5 mg/ kg/h) and remifentanil (0.1 ug/kg/h), and esketamine group was pumped with propofol (5 mg/kg/h) and esketamine (0.5 mg/kg/h). Rocuronium was administered as needed in intermittent boluses of 0.3 mg/kg intraoperatively. After the lateral decubitus position is set up and the paravertebral block (T4 and T6 levels, 0.5% ropivacaine, 10 ml each) was performed under ultrasound guidance, supplemented by 0.75% ropivacaine infiltration at the surgical site upon skin closure. At the completion of the surgery, patients were given 200 mg sugammadex sodium as an antagonistic residual muscle relaxant. They were transferred to the post-anesthesia care unit (PACU) after tracheal extubation and full recovery of consciousness, and returned to the thoracic surgery ward for further treatment after reaching the discharge criteria of PACU. Postoperative analgesia was provided without patient-controlled intravenous analgesia (PCIA). We employed a modified Brice questionnaire to assess the occurrence of intraoperative awareness. The confusion assessment method (CAM) was used to assess postoperative delirium (POD). Rescue analgesia with intravenous flurbiprofen axetil (50 mg) was administered when NRS scores reached ≥4. Rescue antiemetic therapy (intravenous palonosetron 0.075 mg) was provided for postoperative nausea and vomiting (PONV) scores reached ≥4.

Update note (2026-01-04): The record was updated to correct terminology/wording errors (e.g., static vs dynamic compliance; increased intracranial pressure vs intracranial pressure) and to clarify that PCIA was not used. Meanwhlie, a more detailed account that specifies the anesthetic management protocol with greater precision was provided. One prespecified secondary outcome (inflammatory biomarkers) was not collected; therefore, no data are available for that outcome.

ELIGIBILITY:
Inclusion Criteria

1. ASA physical status I-II
2. age 18-70 years
3. thoracoscopic segmentectomy or lobectomy is proposed under general anesthesia due to pulmonary nodule
4. informed consent was obtained Exclusion Criteria

(1) body mass index ˃30 kg/m2 or ˂ 19 kg/m2 (2) preoperative use of opioids, acute and chronic pain or hyperalgesia (3) significant ischemic heart disease, including preoperative coronary artery disease, severe angina, heart failure, or structural heart disease (e.g., significant valvular disease) (4) severe hepatic and renal failure before operation (5) history of mental illness or alcoholism (6) history of alcohol or drug abuse (7) increased intracranial pressure, elevated intraocular pressure, or a diagnosis of glaucoma (8) poorly controlled or untreated hypertension (9) preeclampsia or eclampsia (10) untreated and undertreated hyperthyroidism (11) inability to complete the required rating scales

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-02-04 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Static Lung Compliance | During the operation (at 30 minutes of one-lung ventilation).
  Respiratory parameters displayed on the anesthesia ventilator were recorded during one-lung ventilation. The formula: static lung compliance = tidal volume/platform pressure (Pplat) - positive end expiratory pressure (PEEP) was used to calculate the compliance of the ventilate lung.

SECONDARY OUTCOMES:
Static lung compliance during operation | At the beginning of double lung ventilation, start of one-lung ventilation, and end of surgery.
  Respiratory parameters displayed on the anesthesia ventilator were recorded. Static lung compliance during operation was calculated as: tidal volume / (Pplat - PEEP).
Perioperative pulmonary function | The day before surgery, one day after surgery, two days after surgery, three days after surgery
  Pulmonary function was measured with a portable spirometer, recording forced vital capacity (FVC), forced expiratory volume in one second (FEV1), and the FEV1/FVC ratio.
Blood pressure | At admission, immediately before intubation, immediately after intubation, at the beginning of double lung ventilation, start of one-lung ventilation, 30 min after the start of one-lung ventilation, end of surgery, and on transfer from the PACU.
  Invasive arterial pressure from the monitor.
Heart rate | At admission, immediately before intubation, immediately after intubation, at the beginning of double lung ventilation, start of one-lung ventilation, 30 min after the start of one-lung ventilation, end of surgery, and on transfer from the PACU.
  Heart rate from the monitor.
Blood gas analysis results | At admission, at the beginning of double lung ventilation, one-lung ventilation for 30 minutes, end of surgery, and transfer from the PACU.
  The patient's arterial blood was collected, and the blood gas analyzer was used to determine the human blood H+ concentration and the gas dissolved in the blood (mainly CO2 and O2) to understand the human respiratory function and acid-base balance.
Serum inflammatory factor levels | not collected
  This secondary outcome was prespecified. However, no perioperative blood samples were collected for inflammatory biomarkers (e.g., IL-6, IL-8, TNF-α) in this completed study; therefore, no data are available for this outcome.
cognitive function | The day before surgery, one day after surgery, three days after surgery
  Mini-mental State Examination (MMSE) was used to evaluate the cognitive function of the patients. The total score of the scale was 30, with the lowest score being 0 and the highest 30. A normal person's MMSE score is usually between 27 and 30 points. If the score is lower than 27, it is necessary to be alert to the existence of cognitive impairment. At the same time, according to different levels of education, the classification criteria are also different. For example, illiteracy below 17 points, primary school education below 20 points, secondary school education below 22 points, college education below 23 points, are considered to have cognitive impairment.
Postoperative nausea and vomiting | 30 min after surgery, 6 h after surgery, 24 h after surgery, and 48 h after surgery
  Postoperative nausea and vomiting were evaluated using the "Nausea and Vomiting Numerical Rating Scale", the lowest score being 0 and the highest 10, 0 was no nausea; 1-3 is classified as mild nausea; 4-6 classified as moderate nausea; In addition, regardless of the degree of nausea, patients should also record whether they are accompanied by vomiting. If they are accompanied by vomiting, select Yes; Not accompanied by vomiting, Select No.
Depression and anxiety | The day before surgery, two days after surgery
  Psychological distress was assessed using the Hospital Anxiety and Depression Scale. Scores of 0-7 on each subscale are classified as "normal", 8-10 as "borderline", and 11-21 as "abnormal" (indicating probable clinical significance).
Postoperative pain | 30 min after surgery, 6 h after surgery, 24 h after surgery, and 48 h after surgery
  The patients' postoperative pain was evaluated using the "Pain Numerical Rating Scale", the lowest score was 0, the highest score was 10, 0 indicates no pain; A 10 is the worst pain imaginable. A score of 1 to 3 indicates mild pain that does not affect sleep; A score of 4 to 6 indicates moderate pain and disturbed sleep. A score of 7 to 10 indicates severe pain that severely interferes with sleep.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No